CLINICAL TRIAL: NCT04439058
Title: Preoperative Stellate Ganglion Block Can Cause Enhanced Recovery After Coronary Arteries Bypass Grafting Surgery
Brief Title: Stellate Ganglion Block Can Cause Enhanced Recovery After Coronary Arteries Bypass Grafting Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: wail abdelaal (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, wail abdelaal, assistant professor of anesthesia, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU R3 /2020
Record Dates: First submitted 2020-06-12; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: US machine Mindray M5 (Shenzhen Mindray Bio-Medical Electronics Co., LTD. Shenzhen, China.) with a linear 38-mm high frequency 10-12 MHz transducer), with an imaging depth of 4 cm. A 50-mm short bevel 22-gauge insulated stimulating needle (PAJUNK® GmbH Medizin technologie, Deutschland) was used
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine+lignocaine (Active Comparator): will receive ultrasound guided left stellate ganglion block just after induction of anesthesia with10 ml of bupivacaine 0,25%+ 5ml lignocaine 1%(20 patients).
  Under complete aseptic precautions an ultrasound guided left stellate ganglion block (paratracheal technique ) The patient placed in the supine position with the head in the neutral position and slightly extended.
  The US probe placed at the level of the cricoid cartilage. The transverse process of the sixth cervical vertebra identified by its prominent anterior tubercle. Also, the longus colli muscle and its overlying prevertebral fascia anterior to the C6 vertebral body and deep to the carotid artery. skin infiltration with local anesthetic, the needle inserted from lateral to medial using the in-plane technique. The aim was to inject the local anesthetics deep to the prevertebral fascia and above the longus colli
  Interventions: Other: ultrasound guided left stellate ganglion block
- Normal saline (Other): will receive ultrasound guided left stellate ganglion block just after induction of anesthesia with 15 ml of normal saline (20 patients).
  US machine Mindray M5 (Shenzhen Mindray Bio-Medical Electronics Co., LTD. Shenzhen, China.) with a linear 38-mm high frequency 10-12 MHz transducer), with an imaging depth of 4 cm. A 50-mm short bevel 22-gauge insulated stimulating needle (PAJUNK® GmbH Medizin technologie, Deutschland
  Interventions: Other: ultrasound guided left stellate ganglion block

INTERVENTIONS:
Other: ultrasound guided left stellate ganglion block — Stellate Ganglion Block (SGB) has several established clinical indications Under complete aseptic precautions an ultrasound guided left stellate ganglion block was performed. (paratracheal technique ) ( ) The patient was placed in the supine position with the head in the neutral position and slightly extended. An initial scanning was done with the ultrasound to identify the structures in this area.
  The US probe was placed at the level of the cricoid cartilage. The transverse process of the sixth cervical vertebra was identified by its prominent anterior tubercle. Also, the longus colli muscle and its overlying prevertebral fascia were sought anterior to the C6 vertebral body and deep to the carotid artery. After skin infiltration with local anesthetic, the needle was inserted from lateral to medial using the in-plane technique. The aim was to inject the local anesthetics deep to the prevertebral fascia and above the longus colli

SUMMARY:
The effects of SGB on the cardiovascular system remain controversial since the cardiac sympathetic nerves pass through the stellate ganglion. SGB is expected to have an ameliorative effect on impaired coronary circulation and cardiac function and thus to be well suited to the treatment of angina pectoris and myocardial infarction

DETAILED DESCRIPTION:
investigators chose left SGB being safer with regards conductivity changes when compared to right SGB, in the present study investigators are trying to examine and compare whether coronary reperfusion in patients undergoing coronary artery bypass grafting who were subject to ultrasound guided left Stellate ganglion block (SGB ) performed in the induction of anesthesia could decrease post cardiopulmonary bypass ischemic changes, pulmonary hypertension and right ventricular dysfunction leading to enhanced recovery.

Place of work: Ain shams university hospitals cardiovascular surgery academy, Cairo, Egypt.

Number and selection of participants:

40 participants, 20 in each group (2 groups).

ELIGIBILITY:
Inclusion Criteria:

Ischemic heart disease patients age above 18 years

Exclusion Criteria:

allergy to LA, severe COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
change in heart rate | change in heart rate from base line
  heart rate( bpm )
change in Ejection Fraction | change in Ejection Fraction from base line
  Ejection Fraction(%)
change in blood pressure | change in blood pressure from base line
  MAP, Systemic arterial pressure ( mmHg )
change in cardiac rhythm | change in cardiac rhythm from base line
  incidence of AF or VF(BPM)

SECONDARY OUTCOMES:
effect of preoperative stellate ganglion block on enhanced recovery after coronary arteries bypass grafting surgery | change of troponin level from base line
  measuring troponin level (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: diaa marzouk, M.D, Study Director — professor
Locations (1):
- Wail Abdelaal, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No